CLINICAL TRIAL: NCT00510926
Title: CML/021 "A Phase II Exploratory Study of IMATINIB High Dose (800mg/gg) in the Treatment of Newly Diagnosed Intermediate Risk Chronic Myeloid Leukemia in Chronic Phase"
Brief Title: Exploratory Study of IMATINIB High Dose in Intermediate Risk Chronic Myeloid Leukemia in Chronic Phase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Bologna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CML/021
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2007-08-03 (Estimated); Status verified 2007-08

CONDITIONS: Myeloid Leukemia, Chronic, Chronic-Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesilate (Glivec)

SUMMARY:
Results in CP are better in patients treated early after the onset of the disease with respect to late CP . To date, the early McR rate to imatinib is clearly higher in low and intermediate risk versus high risk (88 and 84% versus 65%). High dose of imatinib, as shown in phase I-III trials may offer the possibility to increase the response rate of patients belonging to this risk category.

DETAILED DESCRIPTION:
This is a phase II multicenter, open-label study designed to investigate the efficacy (hematological response, cytogenetic response and molecular response) and feasibility (tolerance, compliance and safety) of the tyrosine kinase inhibitor imatinib mesylate (formerly STI 571, GLIVECÔ, Novartis Pharma) at high dose (800 mg/daily) (serial number protocol ICSG/CML/021) in patients with Ph+ chronic myeloid leukemia (CML) in chronic phase (CP) previously untreated, at intermediate Sokal risk.

With aIFN, responses (HR and CgR) are significantly influenced by the disease phase and, in CP patients, by risk. aIFN induces rare and short lived HR and CgR (any degree) in late CP and particularly in accelerated and blastic phase.

Moreover, in CP patients Sokal's risk influences significantly the probability of obtaining a MCgR after aIfaIFN . As far as survival, after aIFN even in CCgR patients, the long term survival is signifcantly influenced by risk. The European investigators on Interferon in CML (EICML) collected informations on response and survival on 317 complete cytogenetic responders to IFN. The 10 years survival of the whole patients population was 75% but, after stratification by risk, a significant difference in 10 years survival rates was found in favour of low risk patients (89%) if compared with intermediate risk (70%) and high risk patients (54%) (low vs high risk p 0.0001; intermediate vs high p 0.003, log-rank test).

Long term survival data still lacks after imatinib. However, it has been already shown that the disease phase influences the efficacy of imatinib in CML: responses (HR and particularly CgR) are better in CP versus accelerated and blastic phase. Results in CP are better in patients treated early after the onset of the disease with respect to late CP . To date, the early McR rate to imatinib is clearly higher in low and intermediate risk versus high risk (88 and 84% versus 65%).

Two scoring systems are available for disease risk evaluation, Sokal and Euro. Sokal risk is based on chemotherapy treated patients and Euro risk is based on aIFN trated patients: it is not known to date if one or both of the scoring systems will apply to imatinib treated patients. Moreover, the Sokal system has been applied to stratify the patients by risk in all the large clinical trials of imatinib in CML in the last 3 years and consequently, Sokal score will be employed in the present trial.

Study objectives

Primary:

To determine the rate of complete cytogenetic response at 12 months in adult patients with previously untreated intermediate Sokal risk CML treated with imatinib 800 mg/daily

Secondary:

To determine:

1. The rate of major cytogenetic response at 6 and 12 months.
2. The kinetic of cytogenetic response at 6 and 12 months
3. The duration of complete cytogenetic response.
4. The rate and duration of hematologic response.
5. The degree and the timing of molecular response
6. The time to accelerated and blast crisis and overall survival
7. The safety and tolerability of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age >/=18 years
* First chronic phase, less than 6 months of duration
* Intermediate Sokal's risk
* Ph positive
* No previous treatment or hydroxiurea only.
* Performance status (ECOG/WHO) < or = 2
* Written informed consent

Exclusion Criteria:

* Age <18
* Low or high Sokal risk score.
* More than 6 months from diagnosis.
* Second chronic, accelerated or blastic phase
* Scheduled allogeneic stem cell transplantation within 1 year from diagnosis.
* Performance status (ECOG/WHO) > 2 (see Appendix 2)
* Inability to provide written informed consent
* Pregnancy
* Formal refusal of any recommendation of a safe contraception
* Alcohol or drug addiction
* Altered hepatic or renal function as defined by AST/ALT or bilirubine > 3 times upper normal limits (UNL) and by creatinine ³ 20mg/L Any other disease or condition that by the advise of the responsible physician would make the treatment dangerous for the patient or would make the patient ineligible for the study, including physical, psychiatric, social and behavioural problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2004-01; Study Completion 2006-11

PRIMARY OUTCOMES:
Rate of complete cytogenetic response at 12 months

SECONDARY OUTCOMES:
The rate of major cytogenetic response at 6 and 12 months.
The kinetic of cytogenetic response at 6 and 12 months
The duration of complete cytogenetic response.
The rate and duration of hematologic response.
The degree and the timing of molecular response (see section 13 and 14.5).
The time to accelerated and blast crisis and overall survival (see section 14.2)
The safety and tolerability of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Baccarani, MD, Principal Investigator — Policlinico S.Orsola-Malpighi - Istituto di Ematologia e Oncologia Medica "L. e A.Seràgnoli", Bologna
Locations (1):
- Policlinico S.Orsola-Malpighi, Istituto di Ematologia e Oncologia Medica "L. e A. Seràgnoli", Bologna, Italy

REFERENCES:
- [Derived] Gugliotta G, Castagnetti F, Breccia M, Albano F, Iurlo A, Intermesoli T, Abruzzese E, Levato L, D'Adda M, Pregno P, Cavazzini F, Stagno F, Martino B, La Barba G, Sora F, Tiribelli M, Bigazzi C, Binotto G, Bonifacio M, Caracciolo C, Soverini S, Foa R, Cavo M, Martinelli G, Pane F, Saglio G, Baccarani M, Rosti G; Gruppo Italiano Malattie Ematologiche dell'Adulto - Chronic Myeloid Leukemia Working Party. Incidence of second primary malignancies and related mortality in patients with imatinib-treated chronic myeloid leukemia. Haematologica. 2017 Sep;102(9):1530-1536. doi: 10.3324/haematol.2017.169532. Epub 2017 Jun 1. PMID 28572163
- [Derived] Castagnetti F, Gugliotta G, Baccarani M, Breccia M, Specchia G, Levato L, Abruzzese E, Rossi G, Iurlo A, Martino B, Pregno P, Stagno F, Cuneo A, Bonifacio M, Gobbi M, Russo D, Gozzini A, Tiribelli M, de Vivo A, Alimena G, Cavo M, Martinelli G, Pane F, Saglio G, Rosti G; GIMEMA CML Working Party. Differences among young adults, adults and elderly chronic myeloid leukemia patients. Ann Oncol. 2015 Jan;26(1):185-192. doi: 10.1093/annonc/mdu490. Epub 2014 Oct 30. PMID 25361995
- [Derived] Luatti S, Castagnetti F, Marzocchi G, Baldazzi C, Gugliotta G, Iacobucci I, Specchia G, Zanatta L, Rege-Cambrin G, Mancini M, Abruzzese E, Zaccaria A, Grimoldi MG, Gozzetti A, Ameli G, Capucci MA, Palka G, Bernasconi P, Palandri F, Pane F, Saglio G, Martinelli G, Rosti G, Baccarani M, Testoni N; Gruppo Italiano Malattie Ematologiche dell'Adulto (GIMEMA) Working Party on CML. Additional chromosomal abnormalities in Philadelphia-positive clone: adverse prognostic influence on frontline imatinib therapy: a GIMEMA Working Party on CML analysis. Blood. 2012 Jul 26;120(4):761-7. doi: 10.1182/blood-2011-10-384651. Epub 2012 Jun 12. PMID 22692507
- [Derived] Gugliotta G, Castagnetti F, Palandri F, Breccia M, Intermesoli T, Capucci A, Martino B, Pregno P, Rupoli S, Ferrero D, Gherlinzoni F, Montefusco E, Bocchia M, Tiribelli M, Pierri I, Grifoni F, Marzocchi G, Amabile M, Testoni N, Martinelli G, Alimena G, Pane F, Saglio G, Baccarani M, Rosti G; Gruppo Italiano Malattie Ematologiche dell'Adulto CML Working Party. Frontline imatinib treatment of chronic myeloid leukemia: no impact of age on outcome, a survey by the GIMEMA CML Working Party. Blood. 2011 May 26;117(21):5591-9. doi: 10.1182/blood-2010-12-324228. Epub 2011 Mar 30. PMID 21450900
- [Derived] Marzocchi G, Castagnetti F, Luatti S, Baldazzi C, Stacchini M, Gugliotta G, Amabile M, Specchia G, Sessarego M, Giussani U, Valori L, Discepoli G, Montaldi A, Santoro A, Bonaldi L, Giudici G, Cianciulli AM, Giacobbi F, Palandri F, Pane F, Saglio G, Martinelli G, Baccarani M, Rosti G, Testoni N; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Working Party on Chronic Myeloid Leukemia. Variant Philadelphia translocations: molecular-cytogenetic characterization and prognostic influence on frontline imatinib therapy, a GIMEMA Working Party on CML analysis. Blood. 2011 Jun 23;117(25):6793-800. doi: 10.1182/blood-2011-01-328294. Epub 2011 Mar 29. PMID 21447834
- [Derived] Testoni N, Marzocchi G, Luatti S, Amabile M, Baldazzi C, Stacchini M, Nanni M, Rege-Cambrin G, Giugliano E, Giussani U, Abruzzese E, Kerim S, Grimoldi MG, Gozzetti A, Crescenzi B, Carcassi C, Bernasconi P, Cuneo A, Albano F, Fugazza G, Zaccaria A, Martinelli G, Pane F, Rosti G, Baccarani M. Chronic myeloid leukemia: a prospective comparison of interphase fluorescence in situ hybridization and chromosome banding analysis for the definition of complete cytogenetic response: a study of the GIMEMA CML WP. Blood. 2009 Dec 3;114(24):4939-43. doi: 10.1182/blood-2009-07-229864. Epub 2009 Oct 1. PMID 19797518
- [Derived] Castagnetti F, Palandri F, Amabile M, Testoni N, Luatti S, Soverini S, Iacobucci I, Breccia M, Rege Cambrin G, Stagno F, Specchia G, Galieni P, Iuliano F, Pane F, Saglio G, Alimena G, Martinelli G, Baccarani M, Rosti G; GIMEMA CML Working Party. Results of high-dose imatinib mesylate in intermediate Sokal risk chronic myeloid leukemia patients in early chronic phase: a phase 2 trial of the GIMEMA CML Working Party. Blood. 2009 Apr 9;113(15):3428-34. doi: 10.1182/blood-2007-08-103499. Epub 2009 Feb 11. PMID 19211938